CLINICAL TRIAL: NCT05351801
Title: Proof of Concept Trial of Cannabis Derivatives in Neuropathic Pain
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NURP-002-20F
Record Dates: First submitted 2022-04-08; First posted 2022-04-28 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Diabetic Neuropathic Pain; Peripheral Neuropathic Pain
MeSH Terms: interventions — Dronabinol; nabiximols

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, placebo-controlled, parallel group Phase II study with randomization to one of the four treatment arms: 1) 10 mg mg THC , 2) 800 mg CBD , 3) 10.8 mg THC + 10 mg CBD , and 4) placebo. The 8-week treatment phase comprises a 2-week up-titration, 4 weeks maintenance on the target dose followed by 2 weeks down-titration, to minimize cannabis withdrawal syndrome. The two-weeks up titration phase is to minimize side effects and improve tolerability. Efficacy will be assessed by responses during the 4-week target dose phase.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- THC (Syndros) (Active Comparator): Target dose of 10mg per day.
  Interventions: Drug: THC (Syndros); Drug: Placebo
- CBD (Epidolex) (Active Comparator): Target dose of 800 mg per day.
  Interventions: Drug: CBD (Epidolex); Drug: Placebo
- THC + CBD (Nabiximols) (Active Comparator): Target dose of 10.8 mg / 10 mg per day.
  Interventions: Drug: THC + CBD (Nabiximols); Drug: Placebo
- Placebo (Placebo Comparator): Identical in appearance to the three active comparators.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: THC (Syndros) — Participants will receive a target dose of 10mg per day of THC (Syndros).
  Arms: THC (Syndros)
Drug: CBD (Epidolex) — Participants will receive a target dose of 800 mg per day of CBD (Epidolex).
  Arms: CBD (Epidolex)
Drug: THC + CBD (Nabiximols) — Participants will receive a target dose of 10.8 mg / 10 mg per day of THC + CBD (Nabiximols).
  Arms: THC + CBD (Nabiximols)
Drug: Placebo — Placebo

SUMMARY:
Chronic neuropathic pain (CNP) is disabling. Research on frontline treatments for CNP, shows inconsistent outcomes and dissatisfaction among Veterans. Veterans and clinicians have shown significant interest in cannabis derivatives (THC, CBD) for neuropathic pain control, but there are no well-controlled trials guiding expectations for benefit and adverse outcomes associated with cannabis for CNP. Because Veterans are likely to present with pain and pain-related polymorbidity significantly differing from that of civilians, a well-structured clinical trial of cannabinoids for Veterans with CNP is vital.

DETAILED DESCRIPTION:
Chronic pain is a significant burden to United States Veterans and is a particular concern for Veterans. One of the causes of pain is chronic neuropathic pain (CNP). Frontline treatment for CNP, show inconsistent outcomes and have significant side effects. The ongoing opioid crisis has led to significant interest in safe and effective alternatives for pain control, and there is a significant need for research on desirable options for pain control that are likely to improve treatment adherence and outcomes. Veterans groups and Veterans Affairs clinicians have expressed significant interest in cannabis and its principal constituents (delta-9-tetrahydrocannabinol, THC; cannabidiol, CBD) for pain management, but the extant research describing the potential risks and benefits of cannabis for pain is weak. This randomized trial was developed as a proof of concept study to determine if cannabis constituents (THC, CBD, and THC+CBD) are superior to placebo in reducing pain in Veterans with CNP. The study is to recruit a sample of 320 adult Veterans who meet diagnostic criteria for high-impact CNP, are on stable treatment(s) for CNP, are not current cannabis users and who do not meet diagnostic criteria for Cannabis Use Disorder. This randomized phase II, 4-arm clinical trial aims to determine if cannabis constituents (THC, CBD) or their combination (THC+CBD) are superior to placebo in reducing pain in Veterans with CNP. This trial will offer the first evidence describing the potential benefits and adverse effects of cannabinoids for CNP in Veterans.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written consent
* Veterans 21 years and older at the date of screening
* Meet diagnostic criteria for neuropathic pain as defined by the Neuropathic Pain Special Interest Group of the International Association for the Study of Pain (NeuPSIG)
* Meet criteria for persistent, high-impact pain criteria.
* Presence of allodynia confirmed by one of the screening dynamic brush tests

Exclusion Criteria:

* Peripheral neuropathy is not a primary source of neuropathic pain
* Hypersensitivity to THC, CBD, or THC/CBD
* Self-report of cannabis use during screening phase confirmed by positive urine toxicology for THC-COOH as measured and resulted at visit 5 before randomization
* Unwilling to refrain from using cannabis or cannabis-based products through the entire duration of the study
* Diagnosis of DSM-5 Cannabis Use Disorder in the past 6 months
* Current DSM-5 diagnosis of cannabis use disorder, substance use disorder or serious psychiatric disorders
* Actual change or intent to change is greater than a 20% change (increase or decrease) in any other medication for pain or non-pharmacological treatment from 4 weeks before the screening appointment until completion of study (i.e., visit 13)
* Opioid doses > 400 mg MME (morphine milligram equivalent)
* Women who are pregnant or breastfeeding, or who intend to become pregnant in the 12 weeks from enrollment
* Any current unstable or concerning medical condition that would place the patient at increased risk, including hepatic, respiratory, immunological, cardiovascular, endocrine, or renal disease, or in the opinion of the investigator, prevents adherence with the protocol
* Need for immediate psychiatric hospitalization
* Enrolled in a medical marijuana program
* Federal employee

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2023-06-21 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
To compare the short-term efficacy of THC, CBD, or THC+CBD vs Placebo on Neuropathic Pain as measured by the Numeric Rating Scale of Pain | Baseline, Week 6
  The mean change in the weekly average of daily Numeric Rating Scale (NRS) pain score (0-10 scale; 0=no pain, 10=worst possible pain) from baseline to week 6.

SECONDARY OUTCOMES:
To assess the efficacy of THC, CBD, or THC+CBD vs Placebo in pain quality (allodynia) as measured by the Quantitative Sensory Testing. | Baseline, Week 2, Week 4, Week 6, Week 8
  Allodynia measured by Quantitative Sensory Testing (QST) (0-10 scale; 0=no pain, 10=worst possible pain)
To assess the efficacy of THC, CBD, or THC+CBD vs Placebo in disability and function as measured by the Neuropathic Pain Scale. | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8
  Neuropathic Pain Scale (NPS) total score; 7 different questions/sensations (for each individual item 0-10 scale; 0= not present/no pain, 10= most sensation). Individual scores analyzed separately for pain quality and mean score analyzed for overall neuropathic pain).
To assess the efficacy of THC, CBD, or THC+CBD vs Placebo in disability and function as measured by the Gait Speed Test | Baseline, Week 4, Week 8
  Distance walked (meters)/time (seconds) measured by Gait Speed Test (lower score = worse, higher score =better)
To assess the efficacy of THC, CBD, or THC+CBD vs Placebo in mean changes in perceived improvement as measured by the Patient Global Impression of Change | Baseline, Week 2, Week 4, Week 6, Week 8
  Patient Global Impression of Change (PGIC) 1-7 point ordinal scale assessed (1 = worse, 7 = better)
To assess the efficacy of THC, CBD, or THC+CBD vs Placebo in mean changes in perceived improvement as measured by the patient satisfaction visual analog scale. | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8
  Patient satisfaction with intervention on visual analog scale (VAS, 0-100, 0=no satisfaction, 100 = complete satisfaction).
To assess the efficacy of THC, CBD, or THC+CBD vs Placebo in mean changes in quality of life measured by the Veterans RAND 12 Item Health Survey | Baseline, Week 4, Week 8
  Mental Component Score (MCS) and Physical Component Score (PCS) measured by Veterans RAND 12 Item Health Survey (VR-12). VR-12 is an algorithmic score with ranges from 0-100 (0 indicates worse health-related quality of life and 100 represents better health-related quality of life).
To assess the efficacy of THC, CBD, or THC+CBD vs Placebo in anxiety measured by the Generalized Anxiety Disorder-7. | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8
  Generalized anxiety symptomology is measured by Generalized Anxiety Disorder-7 (GAD-7) total score. (total score ranges from 0-21; Score 0-4 = minimal anxiety, Score 5-9 = mild anxiety, Score 10-14 = moderate anxiety, Score 15-21 = severe anxiety)
To assess the efficacy of THC, CBD, or THC+CBD vs Placebo in pain quality as measured by the Short Form McGill Pain Questionnaire (SF-MPQ-2). | Baseline, Week 2, Week 4, Week 6, Week 8
  Short Form McGill Pain Questionnaire (SF-MPQ-2) total score and four subscales (continuous pain, intermittent pain, predominantly neuropathic pain, affective). (0= no pain to 5= excruciating pain)
To assess the efficacy of THC, CBD, or THC+CBD vs Placebo in mean changes in disability and function as measured by the Brief Pain Inventory-Diabetic Peripheral Neuropathy. | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8
  Brief Pain Inventory-Diabetic Peripheral Neuropathy (BPI-DPN) pain intensity score (first four items 0-10; 10= pain as bad as can imagine) (remaining items 0% (no relief)-100% (complete relief)) and pain interference score (0-10, 10= completely intense).
To assess the efficacy of THC, CBD, or THC+CBD vs Placebo in emotional functioning (severity of depression) as measured by the Patient Health Questionnaire-9. | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8
  Severity of depression is measured by Patient Health Questionnaire-9 (PHQ-9) total score (0-27; 0=none, 27=worst).
To assess the efficacy of THC, CBD, or THC+CBD vs Placebo in emotional functioning (PTSD symptoms) as measured by the PTSD Checklist-DSM-5 (PCL-5). | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8
  PTSD symptoms are assessed by PTSD Checklist-DSM-5 (PCL-5) total score symptom severity score (0-80; 0= not at all to 80= worst).

CONTACTS AND LOCATIONS:
Overall Officials: Deepak D'Souza, MD MBBS, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT; Donald McGeary, PhD, Principal Investigator — South Texas Health Care System, San Antonio, TX
Locations (5):
- United States (5):
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - Providence VA Medical Center, Providence, RI, Providence, Rhode Island
  - South Texas Health Care System, San Antonio, TX, San Antonio, Texas
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No